CLINICAL TRIAL: NCT04585425
Title: God Nat - God Dag. A Randomized Controlled Trial of Bedtime Music as Early Intervention for Sleep-onset Insomnia
Brief Title: Music for Sleep-onset Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University Hospital Heidelberg (Other); University College Nordjylland (Unknown); University of Oxford (Other); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M&I2020
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Treatment as usual including sleep hygiene advice
  Interventions: Behavioral: Sleep hygiene advice
- Intervention (Experimental): Treatment as usual (sleep hygiene advice) and bedtime music listening
  Interventions: Behavioral: Sleep hygiene advice; Behavioral: Bedtime music listening

INTERVENTIONS:
Behavioral: Sleep hygiene advice — Participants receive standard sleep hygiene advice.
Behavioral: Bedtime music listening — Participants in the intervention group listen to their preferred sleep playlist daily at bedtime for minimum 30 minutes.
  Arms: Intervention

SUMMARY:
The study is a randomized controlled trial evaluating the effect of bedtime music as an early intervention for sleep-onset insomnia in adults. The investigators use a randomized controlled trial design with two parallel groups. All participants receive sleep hygiene advice as standard treatment and participants in the intervention group are additionally asked to listen to a sleep playlist daily at bedtime. Subjective and objective sleep measures are evaluated before and after the 4 weeks intervention period. In addition, follow-up measures of subjective outcomes are assessed 4 weeks after the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Sleep-onset insomnia for 3-18 months

Exclusion Criteria:

1. use of medications (benzodiazepines, z-drugs, antidepressive and anti-psychotic drugs)
2. alcohol or substance abuse
3. pregnant or breastfeeding women
4. other sleep disorders (e.g. sleep apnea, restless leg syndrome, etc.)
5. current psychiatric disorder or a history of psychotic disorders
6. somatic disorders interfering with sleep (e.g. critical illness, pain disorders, neuro-degenerative disorders)
7. shift work.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | Change from baseline to after the 4-week intervention period.
  Measured with the Insomnia Severity Index, range 0-28 with higher scores indicating more severe insomnia.

SECONDARY OUTCOMES:
Sleep quality | Change from baseline to after the 4-week intervention period.
  Measured with the Pittsburgh Sleep Quality Index, range 0-21 with higher scores indicating more sleep problems.
Sleep initiation difficulties | Change from baseline to after the 4-week intervention period.
  Difficulties initiating sleep as measured with Pittsburgh Sleep Quality Index subscale
Objective sleep quality | Change from baseline to after the 4-week intervention period.
  Objective sleep quality as measured with polysomnography
Sleep-wake pattern | Change from baseline to after the 4-week intervention period.
  Sleep-wake pattern as measured with wrist-actigraphy
Quality of life | Change from baseline to after the 4-week intervention period.
  Quality of life as measured with SF-36, range 0-100 with higher scores indicating better quality of life.
Pre-sleep arousal | Change from baseline to after the 4-week intervention period.
  Pre-sleep arousal as measured with the Pre-Sleep Arousal Scale, range 8-40 with higher scores indicating higher pre-sleep arousal.

OTHER OUTCOMES:
Depressive symptoms | Change from baseline to after the 4-week intervention period.
  Depressive symptoms as measured with Beck Depression Inventory II, range 0-63 with higher scores indicating more severe depression.
Anxiety | Change from baseline to after the 4-week intervention period.
  Anxiety as measured with the State-Trait Anxiety Inventory, range 0-80 with higher scores indicating more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kira V Jespersen, PhD, Study Director — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jespersen KV, Pando-Naude V, Koenig J, Jennum P, Vuust P. Listening to music for insomnia in adults. Cochrane Database Syst Rev. 2022 Aug 24;8(8):CD010459. doi: 10.1002/14651858.CD010459.pub3. PMID 36000763